CLINICAL TRIAL: NCT01600690
Title: Evaluation of the Effects of 5-day Statin Withdrawal on Endothelial Progenitor Cells and Inflammatory Markers in Type 2 Diabetic Patients. A Controlled Randomized Study
Brief Title: Effects of 5-day Statin Withdrawal on Endothelial Progenitor Cells and Inflammatory Markers in Type 2 Diabetic Patients
Acronym: SStatin-EPC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Gian Paolo Fadini, Assistant Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2616P
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes Mellitus; Atherosclerosis; Dyslipidemia
Keywords: Stem cells; Regeneration; Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis; Dyslipidemias; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continue statin regimen (No Intervention): Patients randomized to this arm will continue their usual statin regimen and dose, without any intervention.
- Statin withdrawal (Experimental): Patients randomized to this arm will stop statin treatment for 5 days.
  Interventions: Other: Statin withdrawal

INTERVENTIONS:
Other: Statin withdrawal — Patients are instructed to stop taking statin pills for the duration of the study. The rest of therapy will remain unchanged.
  Arms: Statin withdrawal

SUMMARY:
Statins are commonly prescribed to lower cardiovascular risk in primary and secondary prevention. Despite their well known efficacy, statin withdrawal is a common event. Even a short term statin withdrawal can have dramatic consequences on atherosclerotic plaque stability, owing to a rebound in cholesterol levels and inflammation.

The effects of a short term statin withdrawal on endothelial progenitor cells (EPC) and monocyte/macrophage polarization is unknown.

In this study, the investigators will explore the effects of a 5-day statin withdrawal on EPC and monocyte/macrophage polarization, together with other inflammatory biomarkers in type 2 diabetic patients. The investigators hypothesize that statin withdrawal determines a reduction in EPC levels and an inflammatory cell polarization.

Patients will be randomized to continue their habitual statin regimen or to withdraw statin. At baseline and 5 days later, blood samples will be collected for experimental measures.

DETAILED DESCRIPTION:
Statins are commonly prescribed to lower cardiovascular risk in primary and secondary prevention. Despite their well known efficacy with relatively low NNTs, statin withdrawal is a common event for several reasons. Patients often stop statin therapies for long or short periods of time. Even a short term statin withdrawal can have dramatic consequences on atherosclerotic plaque stability, owing to a rebound in cholesterol levels and inflammation. Previous studies have demonstrated worsening of inflammation and endothelial function after a short-term statin withdrawal. This may be even more dramatic in patients who are at increased risk of cardiovascular disease, such as diabetic patients.

Endothelial integrity is accomplished through the contribution of circulating endothelial progenitor cells (EPC) which repair the damaged endothelial layer and contribute to cardiovascular health in general. EPC are stimulated by statins, but there is no data on the effect of statin withdrawal on EPCs.

One important aspect of inflammation is the pro- versus anti-inflammatory polarization of circulating monocyte/macrophage (MM) cells. Schematically, MM can exist in 2 different states of activation: the classically activated pro-inflammatory cells (M1) and the alternatively activated anti-inflammatory cells (M2). The balance between these 2 (M1/M2 ratio) reflects the state of MM polarization. The effects of statin withdrawal on MM polarization is unknown.

In this study, we will explore the effects of a 5-day statin withdrawal on EPC and monocyte/macrophage polarization, together with other inflammatory biomarkers (namely high sensitive C-reactive protein) in type 2 diabetic patients. We hypothesise that statin withdrawal determines a reduction in EPC levels and an inflammatory cell polarization.

Patients will be randomized to continue their habitual statin regimen or to withdraw statin. At baseline and 5 days later, blood samples will be collected for experimental measures (EPC, M1, M2 and hsCRP).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Age 35-80
* Males and Females
* eGFR>30 ml/min/1.73 mq
* On statin therapy from at least 6 months
* Minimal statin dosage: Simvastatin 10 mg; Pravastatin 40 mg; Fluvastatin 80 mg; Rosuvastatin 5 mg; Atorvastatin 10 mg.

Exclusion Criteria:

* Type 1 diabetes mellitus
* Age <35 or >80
* Chronic renal failure (eGFR<30 ml/min/1.73 mq)
* Recent (within 1 month) acute diseases or trauma or surgery
* Chronic inflammatory diseases (e.g. rheumatoid arthritis)
* Active cancer
* LDL cholesterol > 160 mg/dL
* Carotid atherosclerosis (>30% stenosis), coronary artery disease, peripheral arterial disease (Leriche stages II-IV)
* On ezetimibe, fibrates, or niacin
* Therapy with EP hormones
* Pregnancy or lactation
* Inability to provide informed consent

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in EPC levels | 5 days
  Change in EPC levels at day 5 versus baseline will be compared between patients who continued taking statins and patients who withdrawed

SECONDARY OUTCOMES:
Change in M1/M2 polarization | 5 days
  Change in monocyte macrophage pro- (M1) versus anti- (M2) inflammatory polarization at day 5 versus baseline will be compared between patients who continued taking statins and patients who withdrawed
Change in hsCRP | 5 days
  Change in high sensitive C-reactive protein levels at day 5 versus baseline will be compared between patients who continued taking statins and patients who withdrawed

CONTACTS AND LOCATIONS:
Overall Officials: Gian Paolo Fadini, M.D., Study Chair — University of Padova
Locations (1):
- University Hospital Diabetes Outpatient Clinic, Padua, Italy